CLINICAL TRIAL: NCT05294094
Title: Learning Diagnostic Skills Online (German: Diagnostik Skills Online Lernen)
Acronym: DiSkO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruhr University of Bochum (Other)
Collaborators: University of Cologne (Other); University of Kaiserslautern-Landau (Other); Philipps Universität Marburg (Unknown)
Responsible Party: Principal Investigator, Ruth von Brachel, Principal Investigator, Ruhr University of Bochum
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 16DHB3010
Record Dates: First submitted 2022-01-17; First posted 2022-03-24 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Diagnosis, Psychiatric
Keywords: clinical interview; blended learning; diagnostic interview
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: intervention group vs. control group
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): blended learning
  Interventions: Behavioral: blended learning
- control group (Active Comparator): Teaching format as usual
  Interventions: Behavioral: teaching format as usual

INTERVENTIONS:
Behavioral: blended learning — The blended learning course consists of two parts. The first part is an online course with case studies and instructional videos providing basic clinical diagnostic knowledge and the ability to conduct structured clinical interviews. In the second part, learners get to discuss the course content with a teacher, practice their interviewing skills with other students and make a transfer to a real face-to-face diagnostic situation with an actor simulating a patient.
  Arms: intervention group
Behavioral: teaching format as usual — The teaching format as usual represents the usual teaching of clinical diagnostic knowledge and the ability to conduct structured clinical interviews. Also in this intervention students also have the opportunity to discuss the course content with a teacher, practice their interviewing skills with other students and conduct a structured interview with an actor simulating a patient.
  Arms: control group

SUMMARY:
Clinical psychologists give diagnoses to their patients everyday and these diagnoses determine if and how these patients will be treated. Misdiagnoses can have severely adverse effects. Therefore, teaching diagnostic skills to clinical psychologists is very important during their undergraduate, graduate and postgraduate training.

One major problem in teaching diagnostics is that there are too few opportunities to practice with real patients due to legal and ethical restrictions. The aim of the DiSkO-project is, therefore, the development and evaluation of a blended learning course to teach diagnostic skills to (future) clinical psychologists.

In order to make the diagnostic training more practical a series of video files of simulated diagnostic interviews will be presented in an online course. These video files will be divided in different segments and presented with questions and automatic feedback. In a second step, learners will make a transfer to a real face-to-face diagnostic situation with an actor simulating a patient.

The DiSkO- course will be evaluated in a randomized-controlled trial at three universities in Germany (Ruhr-University of Bochum, Philipps University of Marburg, University of Cologne). To test whether students are equally good in administering a diagnostic interview after taking the DiSkO-course compared to students who took part in a traditional face-to-face university course a noninferiority-analysis will be conducted. Furthermore, diagnostic knowledge and attitudes toward evidence-based assessment after taking part in DiSkO vs. the face-to-face course will be compared.

The investigators aim at disseminating the open source DiSkO-course to other universities or institutions of tertiary education in Germany with the aim of improving the diagnostic training for students, better prepare them for their clinical practice and thus improve patients' health care in Germany.

ELIGIBILITY:
Inclusion Criteria:

* Psychology bachelor students of a cooperating university (Ruhr-University of Bochum, University of Cologne, Philipps-University of Marburg)

Exclusion Criteria:

* previous participation in a diagnostic seminar

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2022-02-14 (Actual)

PRIMARY OUTCOMES:
Behavioral Measure: Performance in a structured interview | 13 weeks
  Conducting a 15 minute section of a structured interview with a patient played by an actor. This interview is videotaped and then rated by independent evaluators regarding e.g. rules of correct implementation and clincial interviewing skills.

SECONDARY OUTCOMES:
Knowledge Test A | 1 week
  A test of basic clinical diagnostic knowledge developed and previously piloted by the study authors. Using the data from the piloting, two parallel 15-Item versions (A and B) were created, which students answered before and after the intervention.
Knowledge Test B | 14 weeks
  A test of basic clinical diagnostic knowledge developed and previously piloted by the study authors. Using the data from the piloting, two parallel 15-Item versions (A and B) were created, which students answered before and after the intervention.
Münster Questionnaire for the Evaluation of Seminars - revised (MFE-Sr; Thielsch & Hirschfeld, 2010) | 14 weeks
  7-point Likert scale (min.: 1, max.:7)
  The following 6 Items from the MFE-Sr were used:
  Item Number 14: "The content of this course was too difficult for me." Item Number 15: "The pace of teaching was too fast for me." Item Number 16: "The time commitment associated with the course overwhelmed me." Item Number 25: "I learned a lot in this course." Item Number 26: "I would recommend this course to other students."
  Item 14-16: higher values indicate worse outcome, Item 25-26: higher values indicate better outcome
Website-Clarity, Likeability, Informativeness, and Credibility (Web-CLIC; Thielsch & Hirschfeld, 2019) | 14 weeks
  A 12-item questionnaire measuring a users' subjective view on web content, regarding its clarity, likeability, informativeness and credibility. The whole 12-item scale and one additionally created item regarding the credibility ("I completely trusted the content in DiSkO") were used.
  7-point Likert scale (min.: 1, max.:7) higher values indicate better outcome
Brief scale for teaching evaluation (Zumbach, Spinath, Schahn, Friedrich & Kögel, 2007) | 14 weeks
  The following 3 Items were used:
  Item Number 1: "The subject matter was appropriately illustrated (e.g. by examples, visualizations, etc.)." Item Number 2: "The course was clearly structured." Item Number 3: "The learning objectives of the course were clearly defined."
  7-point Likert scale (min.: 1, max.:7) higher values indicate better outcome
Usability Metric for User Experience - Lite (UMUX-Lite; Lewis et al., 2013) | 14 weeks
  A 2-item scale assessing perceived usability.
  7-point Likert scale (min.: 1, max.:7) higher values indicate better outcome
Visual Aesthetics of Websites Inventory - Short (VisAWI-S; Moshagen & Thielsch, 2013) | 14 weeks
  A 4-item scale measuring subjectively perceived aesthetics. The 4-item scale and one additionally created item ("DiSkO is designed to be visually appealing") were used.
  7-point Likert scale (min.: 1, max.:7) higher values indicate better outcome
Overall impression | 14 weeks
  One item using the german school grading system ranging from 1 (very good) to 6 (unsatisfactory):
  "Overall: I give the course an overall grade of ..."
Acceptance of structured interviews questionnaire (Bruchmüller et al., 2011) | 14 weeks
  A 11-item questionnaire measuring the estimated patient satisfaction with structured interviews.
  Item 1:
  visual analogue scale (0-100) higher values indicate better outcome
  Item 2-11:
  4-point Likert scale (min.: 0, max.:3)
  Item 2,3,4,5 and 8 higher values indicate worse outcome Item 6,7,9,10 and 11 higher values indicate better outcome

OTHER OUTCOMES:
Lesson evaluation | After each lesson during the intervention (during week 8-10)
  Each lesson (1-8) of the online part of the blended learning course was evaluated using the following questions:
  "How much time (in minutes) did you spend working on this lesson?" "How concentrated did you work on the content of this lesson?" "I give this lesson an overall grade ..." "Here is space for your feedback on this lesson (e.g. criticism, suggestions, proposals for improvement)"

CONTACTS AND LOCATIONS:
Overall Officials: Ruth E von Brachel, Dr., Principal Investigator — Ruhr-University Bochum
Locations (3):
- Germany (3):
  - Philipps University of Marburg, Marburg, Hesse
  - Ruhr-University Bochum, Bochum, North Rhine-Westphalia
  - University of Cologne, Cologne, North Rhine-Westphalia

IPD SHARING:
Plan to Share IPD: Yes
All anonymized IPD will be shared with the exception of demographic data which, due to rare constellations, entail a risk of deanonymization of individual participants. The IPD will be made available via the Internet database Psychdata (https://www.psychdata.de) of the Leibnitz Center for Psychological Information and Documentation.
Supporting Information: SAP, Analytic Code
Time Frame: The IPD will become available after data analysis (anticipated: September 2022) and will be shared for at least 10 years.
Access Criteria: In order to access the IPD, users must agree to the Data Recipient Agreement and Terms of Use of the internet database Psychdata (https://www.psychdata.de/index.php?main=take&sub=empfang&lang=eng).
  These, among other things, exclude commercial use of the data, protect the interests of the data providers, and ensure the anonymity of the individuals studied.

REFERENCES:
- [Derived] Bonnin G, Krober S, Schneider S, Margraf J, Pflug V, Gerlach AL, Slotta T, Christiansen H, Albrecht B, Chavanon ML, Hirschfeld G, In-Albon T, Thielsch MT, von Brachel R. A Blended Learning Course on the Diagnostics of Mental Disorders: Multicenter Cluster Randomized Noninferiority Trial. J Med Internet Res. 2024 Nov 27;26:e54176. doi: 10.2196/54176. PMID 39602218